CLINICAL TRIAL: NCT01369433
Title: A Rollover Protocol to Allow Continued Access to Tivozanib (AV 951) for Subjects Enrolled in Other Tivozanib Protocols
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of new studies contributing subjects to this study
Sponsor: AVEO Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AV-951-09-901
Record Dates: First submitted 2010-03-04; First posted 2011-06-09 (Estimated); Results first posted 2020-09-01 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Solid Tumors
Keywords: tivozanib
MeSH Terms: interventions — tivozanib; Paclitaxel; temsirolimus; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- tivozanib renal cell carcinoma (RCC) (Experimental): Subjects who participated in a Phase 2 monotherapy study in RCC and showed tolerability and clinical benefit will be allowed access to tivozanib (AV-951).
  Interventions: Drug: Tivozanib
- tivozanib + temsirolimus (Experimental): Subjects who participated in a Phase 1b study and showed tolerability and clinical benefit will be allowed continued access to the tivozanib (AV-951) + temsirolimus combination.
  Interventions: Drug: Tivozanib + temsirolimus
- tivozanib + paclitaxel (Experimental): Subjects who participated in a Phase 1b study and showed tolerability and clinical benefit will be allowed continued access to the tivozanib (AV-951) + paclitaxel combination.
  Interventions: Drug: Tivozanib + paclitaxel
- tivozanib solid tumors - QTC (Experimental): Subjects who participated in a Phase 1 and showed tolerability and clinical benefit will be allowed continued access to the tivozanib (AV-951).
  Interventions: Drug: Tivozanib (AV-951)
- tivozanib + capecitabine (Experimental): After Ph 1b study tolerable to Tivo + Xeloda®
  Interventions: Drug: Tivozanib + capecitabine
- tivozanib Advanced RCC (Experimental): After biomarker study tolerable to Tivo
  Interventions: Drug: Tivo

INTERVENTIONS:
Drug: Tivozanib + paclitaxel — Subjects will continue to receive 0.5 mg, 1.0 mg, or 1.5 mg of tivozanib once daily for 3 weeks beginning on Day 1, followed by 1 week off treatment. On days when paclitaxel and tivozanib (AV-951) are co-administered, tivozanib will be administered immediately following the end of the paclitaxel infusion. All subjects will continue to receive IV paclitaxel 90 mg/m2, administered over 1 hour once a week for 3 weeks, followed by 1 week off.
  Other Names: Tivo (AV-951) + paclitaxel
  Arms: tivozanib + paclitaxel
Drug: Tivozanib + temsirolimus — Subjects will receive 0.5 mg, 1.0 mg or 1.5 mg of tivozanib (AV-951) once daily for 3 weeks, followed by 1 week off. On days when tivozanib (AV-951) and temsirolimus are co-administered, tivozanib (AV-951) will be administered immediately following temsirolimus infusion. Subjects will receive 15 mg or 25 mg temsirolimus IV once weekly.
  Other Names: Tivo (AV-951) + temsirolimus
  Arms: tivozanib + temsirolimus
Drug: Tivozanib — Subjects will receive 1.0 or 1.5 mg tivozanib (AV-951) capsules once daily for 3 weeks, followed by 1 week off.
  Other Names: Tivo (AV951)
  Arms: tivozanib renal cell carcinoma (RCC)
Drug: Tivozanib (AV-951) — Subjects will receive 1.0 or 1.5 mg tivozanib (AV-951) capsules once daily for 3 weeks, followed by 1 week off.
  Other Names: Tivo, (AV-951)
  Arms: tivozanib solid tumors - QTC
Drug: Tivozanib + capecitabine — Subjects will receive 1.5 mg of tivozanib once daily for 2 weeks beginning on Day 1, followed by 1 week off. Subjects will receive Capecitabine (Xeloda®) 825 mg/m2 or 1000 mg/m² or 1250 mg/m² oral twice daily. Subjects will receive capecitabine twice daily for 2 weeks beginning on Day 1, followed by 1 week off.
  Other Names: Tivo, (AV-951) + capecitabine
  Arms: tivozanib + capecitabine
Drug: Tivo — Subjects will receive 1.5 mg tivozanib once daily beginning on Day 1 for 3 weeks followed by 1 week off treatment.
  Other Names: Tivo, (AV-951)
  Arms: tivozanib Advanced RCC

SUMMARY:
Open-label, multi-center, multi-national rollover study to allow continued access to tivozanib for subjects who have participated in other tivozanib (monotherapy or combination) protocols. Eligible subjects will continue to receive tivozanib at the same dose and schedule as per the original (parent) protocol. The length of time that a subject must be on the parent protocol before rolling over to this protocol will be dictated by the (original) parent protocol. Subjects will be seen by the investigator every 4 weeks (± 5 days). Adverse events and blood pressure will be recorded. At the beginning of Cycle 1 and at the beginning of every odd-numbered cycle (Cycle 3, Cycle 5, etc), clinical laboratory values will be recorded. CT scans to assess disease will be performed at the end of even-numbered cycles (Cycle 2, Cycle 4, etc).

DETAILED DESCRIPTION:
This is an open-label multi-center, multi-national rollover protocol to allow continued access to tivozanib for subjects who have participated in other tivozanib (monotherapy or combination) protocols, who are tolerating study drug, and displaying clinical benefit.

Enrollment to this protocol will remain open to subjects who participate in current and future protocols with tivozanib. The end of the study is the last treatment visit of the last subject at the last site. Enrollment in this protocol will continue until tivozanib becomes commercially available in the country where the subject is being treated. If a subject is experiencing clinical benefit from tivozanib when the study is discontinued, the sponsor will make every effort to assist the subject in obtaining commercially available tivozanib.

This rollover protocol will be open to eligible subjects on current and future protocols with tivozanib. The number of subjects who will enroll is dependent upon the number of subjects enrolled in tivozanib protocols that tolerate the drug, display clinical benefits, and are willing to participate.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must have received tivozanib while enrolled in another protocol, must be tolerating study drug and must currently display clinical benefit. The length of time that a subject must be on the parent protocol before rolling over to this protocol will be dictated by the parent protocol.
2. If female and of childbearing potential, documentation of negative pregnancy test prior to enrollment.
3. Ability to give written informed consent.

Exclusion Criteria:

1. > 4 weeks since discontinuation of tivozanib treatment on a previous protocol
2. If female, pregnant or lactating
3. Sexually active male and pre-menopausal female subjects (and their partners) unless they agree to use adequate contraceptive measures, while on study and for 30 days after the last dose of study drug. All fertile male and female subjects (and their partners) must agree to use a highly effective method of contraception. Highly effective birth control includes (a) intrauterine device plus one barrier method; or (b) 2 barrier methods. Effective barrier methods are male or female condoms, diaphragms, and spermicides (creams or gels that contain a chemical to kill sperm). (Note: Oral, implantable, or injectable contraceptives may be affected by cytochrome P450 interactions, and are not considered effective for this study.)
4. Uncontrolled hypertension: systolic blood pressure > 140 mmHg or diastolic blood pressure >90 mmHg on 2 or more antihypertensive medications, documented on 2 consecutive measurements taken at least 24 hours apart.
5. Newly identified central nervous system (CNS) malignancies or documented progression of CNS metastases; subjects will be allowed only if the CNS metastases have been adequately treated with radiotherapy or surgery. For subjects receiving steroid therapy please refer to Section 6.3 for allowed steroid maintenance therapy.
6. Unhealed wounds (including active peptic ulcers)
7. Serious/active infection or infection requiring parenteral antibiotics
8. Life-threatening illness or organ system dysfunction compromising safety evaluation
9. Psychiatric disorder, altered mental status precluding informed consent or necessary testing
10. Inability to comply with protocol requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2010-06; Primary Completion 2015-06 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Berkenblit, MD, Study Director — AVEO Pharmaceuticals, Inc.
Locations (49):
- United States (27):
  - Translational Genomics Research Institute (TGEN), Scottsdale, Arizona
  - Institute of Urologic Oncology, Los Angeles, California
  - Stanford University, Stanford, California
  - Aurora, Colorado
  - Florida Cancer Specialists, Fort Myers, Florida
  - H. Lee Moffitt Cancer Center & Research Institute Hospital, Inc, Tampa, Florida
  - Beech Grove, Indiana
  - Horizon Oncology Research, Inc., Lafayette, Indiana
  - Wichita, Kansas
  - Medical Oncology LLC, Baton Rouge, Louisiana
  - Jayne Gurtler MD, Laura Brinz MD, Angelo Russo MD and Janet Burroff MD APMC, Metairie, Louisiana
  - Associates in Oncology/Hematology, Rockville, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Grand Rapids, Michigan
  - Tupelo, Mississippi
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Las Vegas, Nevada
  - Lebanon, New Hampshire
  - Chapel Hill, North Carolina
  - Columbus, Ohio
  - The OU Cancer Institute, Oklahoma City, Oklahoma
  - Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute (SCRI), Nashville, Tennessee
  - Austin, Texas
  - Coastal Bend Cancer Center, Corpus Christi, Texas
  - Dallas, Texas
  - Tacoma, Washington
- Canada (3):
  - Hamilton, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
- India (2):
  - AVEO Investigational Site, Madurai
  - AVEO Investigational Site, Mumbai
- Rotterdam, Netherlands
- Russia (11):
  - AVEO Investigational Site, Krasnodar
  - AVEO Investigational Site - Moscow 1, Moscow
  - AVEO Investigational Site - Moscow 2, Moscow
  - AVEO Investigational Site - Moscow 3, Moscow
  - AVEO Investigational Site - Moscow 4, Moscow
  - AVEO Investigational Site - Moscow 5, Moscow
  - AVEO Investigational Site, Obninsk
  - AVEO Investigational Site, Rostov
  - AVEO Investigational Site, Saint Petersburg
  - Stavropol
  - AVEO Investigational Site, Ufa
- Ukraine (5):
  - AVEO Investigational Site, Dnipropetrovsk
  - AVEO Investigational Site, Donetsk
  - AVEO Investigational Site, Kharkiv
  - AVEO Investigational Site, Lviv
  - AVEO Investigational Site, Zaporizhya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Aveo Pharmaceuticals, Inc. official web page — http://www.aveooncology.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects who met all the inclusion and none of the exclusion criteria were enrolled in the study.
Pre-assignment Details: All subjects underwent inclusion and exclusion criteria assessment and all eligible subjects signed the informed consent before undergoing any study related procedures.
  All the study assessments were performed as per the schedule of assessment.
Groups:
- Monotherapy: Subjects received oral tivozanib hydrochloride at the same dose and schedule as during the parent protocol. Studies under monotherapy were AV-951-10-112, AV-951-07-201, AV-951-110-202, AV-951-12-205, and AV-951-09-902. Drug: Tivozanib hydrochloride.
- Combination Therapy: Subjects who were receiving tivozanib hydrochloride combination, continued the combination therapy, as long as it was tolerated, at the same dose and schedule as in the parent protocol. Eligible subjects who received sorafenib in Parent Study AV-951-09-902 at the time of study termination and who rolled into Study AV-951-09-901 began tivozanib hydrochloride at a dose of 1.5 mg/day. Studies under combination therapy were AV-951-07-102, AV-951-07-103, AV-951-08-104, AV-951-10-114, and AV-951-12-204. Combination Drugs: Tivozanib hydrochloride + temsirolimus, Tivozanib hydrochloride + paclitaxel, and Tivozanib hydrochloride + capecitabine.
Period: Overall Study
Arm/Group | Monotherapy | Combination Therapy
Started | 209 | 16
Completed | 0 | 0
Not Completed | 209 | 16
Not completed — Adverse Event | 31 | 1
Not completed — Required significant surgical procedure | 1 | 0
Not completed — Non-compliance | 1 | 0
Not completed — Withdrawal by Subject | 5 | 2
Not completed — Study terminated by Sponsor | 67 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Death | 5 | 0
Not completed — Investigator discretion | 6 | 1
Not completed — Progressive Disease | 92 | 12

BASELINE CHARACTERISTICS:
Population: Of the 225 subjects, 209 subjects had monotherapy treatment during their parent study; the remaining subjects (N=16) had combination therapy
  * Monotherapy: Studies AV-951-10-112, AV-951-07-201, AV-951-110-202, AV-951-12-205, AV-951-09-902.
  * Combination: Studies AV-951-07-102, AV-951-07-103, AV-951-08-104, AV-951-10-114, AV-951-12-204.
Groups:
- Monotherapy: Participants received oral tivozanib hydrochloride at the same dose and schedule as during the parent protocol. Studies under monotherapy were AV-951-10-112, AV-951-07-201, AV-951-110-202, AV-951-12-205, and AV-951-09-902. Drug: Tivozanib hydrochloride.
- Combination Therapy: Participants who were receiving tivozanib hydrochloride combination, continued the combination therapy, as long as it was tolerated, at the same dose and schedule as in the parent protocol. Eligible participants who received sorafenib in Parent Study AV-951-09-902 at the time of study termination and who rolled into Study AV-951-09-901 began tivozanib hydrochloride at a dose of 1.5 mg/day. Studies under combination therapy were AV-951-07-102, AV-951-07-103, AV-951-08-104, AV-951-10-114, and AV-951-12-204. Combination Drugs: Tivozanib hydrochloride + temsirolimus, Tivozanib hydrochloride + paclitaxel, and Tivozanib hydrochloride + capecitabine.
- Total: Total of all reporting groups
Arm/Group | Monotherapy | Combination Therapy | Total
Number analyzed (Participants) | 209 | 16 | 225
Age, Customized [Number; unit: participants]
  18 to >= 75 years | 209 | 16 | 225
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 6 | 86
  Male | 129 | 10 | 139
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 0 | 5
  White | 199 | 16 | 215
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Adverse Events (AEs) and Serious AEs
Description: Safety and tolerability will be assessed in accordance to the protocol of the parent study in which the subjects had participated, before enrolling in the AV-951-09-901 rollover study.
Time Frame: 24 Months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Monotherapy | Combination Therapy
Number analyzed (Participants) | 209 | 16
Participants
  AEs | 178 | 16
  Treatment-related AEs | 159 | 15
  AEs ≥Grade 3 toxicity | 111 | 12
  AEs-study drug interruption | 54 | 6
  AEs-study drug dose reduction | 13 | 0
  AEs-discontinuation of study drug | 31 | 1
  AEs-death | 13 | 1
  Serious Adverse events (SAEs) | 44 | 5
  SAEs ≥Grade 3 toxicity | 38 | 5
  Serious treatment-related AEs | 16 | 0

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Monotherapy | Combination Therapy
Serious Adverse Events (participants affected / at risk) | 44/209 | 5/16
Other Adverse Events (participants affected / at risk) | 178/209 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Monotherapy (N=209) | Combination Therapy (N=16)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 5 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Periproctitis (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Disease progression (General disorders) | 1 | 1
Fatigue (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Pneumonia (Infections and infestations) | 3 | 0
Cystitis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 7 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypochloraemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Spinal cord compression (Nervous system disorders) | 2 | 0
Balance disorder (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0
Dysarthria (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Monotherapy (N=209) | Combination Therapy (N=16)
Anaemia (Blood and lymphatic system disorders) | 11 | 2
Hypothyroidism (Endocrine disorders) | 36 | 3
Diarrhoea (Gastrointestinal disorders) | 87 | 8
Nausea (Gastrointestinal disorders) | 53 | 8
Vomiting (Gastrointestinal disorders) | 28 | 5
Stomatitis (Gastrointestinal disorders) | 25 | 5
Abdominal pain (Gastrointestinal disorders) | 25 | 4
Constipation (Gastrointestinal disorders) | 25 | 3
Dyspepsia (Gastrointestinal disorders) | 25 | 3
Abdominal pain upper (Gastrointestinal disorders) | 17 | 1
Dry mouth (Gastrointestinal disorders) | 15 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 13 | 0
Fatigue (General disorders) | 81 | 13
Oedema peripheral (General disorders) | 17 | 5
Asthenia (General disorders) | 19 | 2
Pain (General disorders) | 15 | 1
Non-cardiac chest pain (General disorders) | 12 | 1
Upper respiratory tract infection (Infections and infestations) | 16 | 0
Urinary tract infection (Infections and infestations) | 13 | 3
Decreased appetite (Metabolism and nutrition disorders) | 48 | 6
Dehydration (Metabolism and nutrition disorders) | 14 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 14 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 11 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 31 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 27 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 27 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 13 | 4
Headache (Nervous system disorders) | 43 | 4
Dizziness (Nervous system disorders) | 25 | 2
Dysgeusia (Nervous system disorders) | 14 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 8 | 6
Anxiety (Psychiatric disorders) | 18 | 2
Insomnia (Psychiatric disorders) | 16 | 2
Depression (Psychiatric disorders) | 11 | 2
Proteinuria (Renal and urinary disorders) | 18 | 3
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 51 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 28 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 26 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 19 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 26 | 5
Dry skin (Skin and subcutaneous tissue disorders) | 9 | 3
Hypertension (Vascular disorders) | 88 | 8
Weight decreased (Investigations) | 31 | 3
Neutropenia (Blood and lymphatic system disorders) | 2 | 2
Leukopenia (Blood and lymphatic system disorders) | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 4
Atrial fibrillation (Cardiac disorders) | 1 | 1
Atrioventricular block first degree (Cardiac disorders) | 0 | 1
Cataract (Eye disorders) | 3 | 1
Lacrimation increased (Eye disorders) | 2 | 2
Eye swelling (Eye disorders) | 0 | 1
Visual impairment (Eye disorders) | 0 | 1
Oral pain (Gastrointestinal disorders) | 11 | 0
Abdominal distension (Gastrointestinal disorders) | 7 | 1
Pancreatitis (Gastrointestinal disorders) | 3 | 1
Toothache (Gastrointestinal disorders) | 3 | 2
Epigastric discomfort (Gastrointestinal disorders) | 0 | 2
Haematochezia (Gastrointestinal disorders) | 1 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 1
Tongue ulceration (Gastrointestinal disorders) | 1 | 1
Abdominal mass (Gastrointestinal disorders) | 0 | 1
Abdominal tenderness (Gastrointestinal disorders) | 0 | 1
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 | 1
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 3 | 1
Malaise (General disorders) | 2 | 1
Disease progression (General disorders) | 1 | 1
Early satiety (General disorders) | 0 | 1
Impaired healing (General disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 2 | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 2
Bile duct obstruction (Hepatobiliary disorders) | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 1
Gallbladder enlargement (Hepatobiliary disorders) | 0 | 1
Nasopharyngitis (Infections and infestations) | 8 | 1
Oral herpes (Infections and infestations) | 3 | 1
Cellulitis (Infections and infestations) | 2 | 1
Folliculitis (Infections and infestations) | 2 | 1
Lung infection (Infections and infestations) | 0 | 1
Liver abscess (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Infected cyst (Infections and infestations) | 0 | 1
Tinea cruris (Infections and infestations) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 3 | 1
Lipase increased (Investigations) | 9 | 1
Blood thyroid stimulating hormone increased (Investigations) | 5 | 2
Prothrombin time prolonged (Investigations) | 0 | 4
International normalised ratio increased (Investigations) | 0 | 3
Neutrophil count decreased (Investigations) | 2 | 1
Blood bilirubin increased (Investigations) | 0 | 2
Low density lipoprotein increased (Investigations) | 1 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1
Alanine aminotransferase decreased (Investigations) | 0 | 1
Aspartate aminotransferase decreased (Investigations) | 0 | 1
Blood bilirubin unconjugated increased (Investigations) | 0 | 1
Blood uric acid increased (Investigations) | 0 | 1
Carbon dioxide increased (Investigations) | 0 | 1
Liver function test abnormal (Investigations) | 0 | 1
Protein total decreased (Investigations) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 4 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 9 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 10 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 1
Dizziness postural (Nervous system disorders) | 4 | 1
Paraesthesia (Nervous system disorders) | 3 | 1
Hyperaesthesia (Nervous system disorders) | 1 | 1
Burning sensation (Nervous system disorders) | 0 | 1
Peroneal nerve palsy (Nervous system disorders) | 0 | 1
Vocal cord paralysis (Nervous system disorders) | 0 | 1
Withdrawal syndrome (Psychiatric disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 5 | 1
Nocturia (Renal and urinary disorders) | 1 | 2
Renal failure (Renal and urinary disorders) | 0 | 2
Renal impairment (Renal and urinary disorders) | 0 | 1
Urethral atrophy (Renal and urinary disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Breast mass (Reproductive system and breast disorders) | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Choking sensation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 2
Rash (Skin and subcutaneous tissue disorders) | 9 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 7 | 2
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 5
Rash pruritic (Skin and subcutaneous tissue disorders) | 3 | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 2 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 2 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 1 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1
Neurodermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 2 | 1
Flushing (Vascular disorders) | 2 | 1
Vena cava thrombosis (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No